CLINICAL TRIAL: NCT05851079
Title: Accurate Screening and Prevention of Cervical Lesions-- Development of Accurate Screening Methods for Cervical Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Wuhan Central Hospital (Other); Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20210333-R
Record Dates: First submitted 2023-04-24; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2/3; Cervical Lesion
Keywords: Screening methods; Cervical Lesion; Sensitivity; Accuracy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Cervical exfoliated cells；Cervical biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1. Stratified experimental design: Relying on the project's clinical multicenter to recruit patients for routine HPV screening in hospital outpatient clinics, for HPV high-risk type-positive subjects. The subjects with positive HPV types will continue to undergo TCT and colposcopic biopsy, and the remaining specimens after routine screening will be collected for high-throughput HPV typing and integrated assays. The sensitivity and accuracy of high-throughput HPV typing and integrated assays were compared with conventional screening methods.
  Interventions: Diagnostic Test: TCT test; Diagnostic Test: Vaginoscopy; Diagnostic Test: High throughput HPV typing and integration detection methods; Diagnostic Test: Cobas HPV test
- 2. Parallel experimental design: A multicenter cohort of 12,000 permanent residents was recruited for routine cervical cancer screening(HPV+TCT combined screening), and the remaining specimens were collected after the conventional screening to test the indexes of high-throughput HPV typing and integrated assays. The sensitivity and accuracy of high-throughput HPV typing and integrated assays were compared with conventional screening methods.
  Interventions: Diagnostic Test: TCT test; Diagnostic Test: High throughput HPV typing and integration detection methods; Diagnostic Test: Cobas HPV test
- 3. Prospective cohort study design:: Based on a multicenter cohort of cervical cancer screening based on the project group, 3000 cervical cancer patients with HPV-positive routine screening and colposcopic biopsies were enrolled. The cohort was followed up regularly for 3 years with routine HPV+TCT and colposcopy, and cervical biopsy if necessary. And specimens remaining after routine screening will be collected for testing of high-throughput HPV typing and integrated assays.
  Interventions: Diagnostic Test: TCT test; Diagnostic Test: Vaginoscopy; Diagnostic Test: High throughput HPV typing and integration detection methods; Diagnostic Test: Cobas HPV test

INTERVENTIONS:
Diagnostic Test: TCT test — These tests were performed on cervical exfoliated cells.
Diagnostic Test: Vaginoscopy — To obtain the results of the patient's pathology report.
  Groups: 1. Stratified experimental design; 3. Prospective cohort study design:
Diagnostic Test: High throughput HPV typing and integration detection methods — This is screening for ≥ cervical intraepithelial tumors (CIN2 or CIN3).
Diagnostic Test: Cobas HPV test — To obtain HPV typing results.

SUMMARY:
The goal of this observational study is to compare the accuracy and sensitivity of High-throughput human papilloma virus(HPV) typing and integrated assays with routine screening protocols (Cobas HPV test combined with thinprep cytologic test(TCT) for the detection of cervical intraepithelial neoplasia in the general and hospital populations.

The main questions it aims to answer are:

* High-throughput HPV typing and integrated assays can screen for ≥ cervical intraepithelial neoplasia (CIN2 or CIN3) with high sensitivity and accuracy.
* High-throughput HPV typing and integrated assays can be promoted as a screening tool for cervical cancer.

Participants will be screened with routine screening protocols (Cobas HPV test combined with TCT test), and if the results are abnormal, colposcopy and cervical biopsy will be performed.

DETAILED DESCRIPTION:
1. Stratified experimental design:

   Relying on the project's clinical multicenter to recruit patients for routine HPV screening in hospital outpatient clinics, for HPV high-risk type-positive subjects. The subjects with positive HPV types will continue to undergo TCT and colposcopic biopsy, and the remaining specimens after routine screening will be collected for high-throughput HPV typing and integrated assays. The sensitivity and accuracy of high-throughput HPV typing and integrated assays were compared with conventional screening methods.
2. Parallel experimental design:

   A multicenter cohort of 12,000 permanent residents was recruited for routine cervical cancer screening(HPV+TCT combined screening), and the remaining specimens were collected after the conventional screening to test the indexes of high-throughput HPV typing and integrated assays. The sensitivity and accuracy of high-throughput HPV typing and integrated assays were compared with conventional screening methods.
3. Prospective cohort study design:

Based on a multicenter cohort of cervical cancer screening based on the project group, 3000 cervical cancer patients with HPV-positive routine screening and colposcopic biopsies were enrolled. The cohort was followed up regularly for 3 years with routine HPV+TCT and colposcopy, and cervical biopsy if necessary. And specimens remaining after routine screening will be collected for testing of high-throughput HPV typing and integrated assays.

4.subject selection:

1. .Stratified study design subjects were selected from patients who were first screened for cervical cancer in hospital outpatient clinics.
2. .Parallel trial design subjects were selected from resident female residents in a cohort of cervical cancer screening established by a clinical center.
3. .The prospective cohort study was designed to include HPV-positive patients in the cohort of cervical cancer screening established by the clinical center and whose cervical lesions were excluded by colposcopic biopsy.

5.This project is a multicenter prospective cohort study to investigate the immediate, 1st year, 2nd year and 3rd year cumulative risk of developing CIN2+ and CIN3+ in HPV 16 or 18-positive patients with positive and negative test results by integrating test results through a logistic Weibull model to assess whether colposcopy can be delayed and thus serve as a cervical cancer screening triage by comparing with risk values and clinical thresholds in the 2019 American Society for Colposcopy and Cervical Pathology(ASCCP)guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. First screening.
2. History of sexual intercourse.

Exclusion Criteria:

1. Previous CIN, cervical cancer or other cervical lesions;
2. History of cervical treatment;
3. Age <25, >70 years;
4. Pregnancy.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Subjects were recruited in the general and hospital populations.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
the risk of cervical intraepithelial neoplasia(CIN) 2 or worse | 3 years
  Patients who meet the requirements for referral colposcopy were further examined for CIN2+ by pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wang, PhD, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's hospital school of medicine zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No